CLINICAL TRIAL: NCT05771571
Title: Acute Effect of a Novel, Functional Olive Oil, Enhanced With Orange Peel Extract, on Postprandial Biomarkers of Inflammation and Oxidative Stress of Volunteers at High Cardiometabolic Risk
Brief Title: Investigation of the Acute Effect of Novel Olive Oil on Postprandial Oxidative Stress Biomarkers (BioliveCT)
Acronym: BioliveCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Aegean (Other)
Responsible Party: Principal Investigator, ANTONIOS KOUTELIDAKIS, Professor of Human Nutrition, University of the Aegean
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Bio622
Record Dates: First submitted 2023-03-03; First posted 2023-03-16 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Cardiometabolic Risk
Keywords: Novel olive oil; Orange peel extract; Postprandial bioactivity; Cardiometabolic risk

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into control and interventional group. In the first study period, the control group consumed the meal with the refined olive oil and the interventional group received the meal with the novel, functional olive oil, enhanced with 10% w/w orange peel extract. After a washout week participants were crossed over and consumed the meals in reverse.
Who Masked: Participant
Masking Description: Only researchers knew the type of the meal consumed by each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The meal contained mashed potatoes, homogenized with refined olive oil.
  Interventions: Other: Control
- Interventional (Other): The meal contained mashed potatoes, homogenized with the functional olive oil, enhanced with orange peel extract
  Interventions: Other: Functional olive oil, enhanced with orange peel extract

INTERVENTIONS:
Other: Functional olive oil, enhanced with orange peel extract — The functional olive oil was enriched with 10% w/w orange peel extract
  Arms: Interventional
Other: Control — Refined olive oil
  Arms: Control

SUMMARY:
The purpose of this study was the investigation of the hypothesis that the enhancement of a refined olive oil with orange peel extract, may improve the postprandial lipidemic, glycemic profile and blood oxidative status, of volunteers with high cardiometabolic risk, due to increased content of bioactive compounds (polyphenols, carotenoids etc.).

DETAILED DESCRIPTION:
In a randomized, acute, single-blinded and cross-over study, participated 21 volunteers with high cardiometabolic risk, aged 30-65, were randomized and divided into two groups. The first group consumed a meal of mashed potatoes with added refined olive oil, rich in fat and carbohydrates (300g, control meal), while the second group consumed mashed potatoes with added olive oil, enhanced with 10% w/w orange peel extract (functional meal). After a one-week washout period, the volunteers were crossed over and consumed the meals in reverse. Blood samples were withdrawn in a fasting state, 30, 90 and 180 min after meal consumption. Plasma Total Antioxidant Capacity (FRAP), serum lipid levels [Total, High-Density Lipoprotein (HDL-) and Low-Density Lipoprotein (LDL-) cholesterol and triglycerides], glucose and uric acid were determined at each time point using a biochemical analyzer (Roche Cobas c111).

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 65 years
* Completion of at least 3 of the following parameters:

  * Hypertension (Systolic pressure ≥ 140mm Hydrargyrum or diastolic pressure ≥ 90mm Hydrargyrum or taking antihypertensive treatment)
  * High levels of LDL-cholesterol (≥130mg/dL)
  * High serum triglycerides (≥150mg/dL)
  * Waist circumference >102cm for men and >98cm for women
  * Family history (Myocardial infarction or sudden death in a 1st degree relative <55 years old)
  * High fasting glucose (100-125 mg/dL)

Exclusion Criteria:

* Diabetes or antidiabetic treatment
* Age <45 and >65 years
* Malignancies
* Liver disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Changes of Antioxidant activity from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Plasma Total Antioxidant Capacity concentration
Changes of Low Density Lipoprotein cholesterol (LDL-cholesterol) from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum LDL-cholesterol concentration

SECONDARY OUTCOMES:
Changes of Total cholesterol from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum total cholesterol concentration
Changes of High Density Lipoprotein Cholesterol (HDL-cholesterol) from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum HDL-cholesterol (HDL-cholesterol) concentration
Changes of glucose from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum glucose concentration
Changes of triglycerides from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum triglycerides concentration
Changes of uric acid from baseline to 30 minutes, 1.5 hours and 3 hours | 3 hours
  Serum Uric Acid concentration

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Aegean, Myrina, Greece

IPD SHARING:
Plan to Share IPD: No
No one individual participant data is planned to be shared.